CLINICAL TRIAL: NCT00460564
Title: A Multicenter Study to Evaluate the Efficacy and Safety in Patients With Post-Stroke Upper Limb Spasticity Receiving a Double-Blind, Placebo-Controlled GSK1358820 Treatment Followed by an Open-Label GSK1358820 Treatment
Brief Title: Study Of GSK1358820 In Patients With Post-Stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTX108509
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Post-Stroke Spasticity; Cerebrovascular Accident
Keywords: Spasticity; Post-Stroke; botulinum toxin type A; Upper Limb
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High-Dose BTX (Active Comparator)
  Interventions: Drug: GSK1358820
- High-Dose Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Low-Dose BTX (Active Comparator)
  Interventions: Drug: GSK1358820
- Low-Dose Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1358820 — botulinum toxin type A
  Arms: High-Dose BTX; Low-Dose BTX
Drug: Placebo — Placebo
  Arms: High-Dose Placebo; Low-Dose Placebo

SUMMARY:
This is a study to confirm the superior efficacy of a single treatment of GSK1358820 over placebo in patients with post-stroke upper limb spasticity of both the wrist and finger flexors using the Modified Ashworth Scale (MAS) wrist score.

DETAILED DESCRIPTION:
This is a study to confirm the superior efficacy of a single treatment of GSK1358820 over placebo in patients with post-stroke upper limb spasticity of both the wrist and finger flexors using the Modified Ashworth Scale (MAS) wrist score.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria:

* Patients with upper limb spasticity who are at least 6 months post stroke and present with spasticity of both the wrist and fingers at the start of double-blind phase (Visit 2).
* Wrist flexor muscle tone of ≥3 and finger flexor muscle tone of ≥2 on the MAS, and at least one functional disability item (i.e., hygiene, pain, dressing or limb posture) with a rating of ≥2 on the Disabilty Assessment Scale (DAS) at the start of double-blind phase (Visit 2).
* Male or female between 20 and 80 years of age at the time of informed consent. For males, only those who can practice contraception during the study period are eligible.
* ≥40kg in weight at the start of double-blind phase (Visit 2).
* Inpatient or outpatient; however, the hospitalization status must remain unchanged during the double-blind phase.
* Written informed consent from the subject him/herself. If the subject's signature is not legible, the attendance of a witness is required.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Bilateral hemiplegia or quadriplegia.
* Presence of fixed contractures of the wrist and/or fingers (absence of range of motion).
* Profound atrophy of the muscles to be injected.
* Previous surgical intervention, phenol block, ethanol block, or muscle afferent block (MAB) for wrist and/or finger spasticity.
* Casting of the study upper limb within 3 months prior to the start of double-blind phase (Visit 2).
* Current treatment with intrathecal baclofen.
* Use of peripheral muscle relaxants (dantrolene sodium, suxamethonium chloride, pancuronium bromide, vecuronium bromide, rocuronium bromide).
* Concurrent use of antibiotics that interfere with neuromuscular transmission, such as aminoglycoside antibiotics (e.g., streptomycin sulfate, kanamycin sulfate, gentamicin sulfate, neomycin sulphate, spectinomycin hydrochloride), polypeptide antibiotics (e.g., polymixin B sulfate), lincomycin antibiotics (e.g., lincomycin hydrochloride, clindamycin), and enviomycin sulfate.
* Previous botulinum toxin therapy.
* Diagnosis of systemic neuromuscular disorders (e.g., myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis).
* Females who are pregnant, nursing, may be pregnant, or planning a pregnancy during the study period.
* Known allergy or hypersensitivity to any ingredient of study medication (e.g., human serum albumin).
* Presence of psychiatric disorder or impairment of intellectual function that may interfere with the subject's ability to give informed consent or the conduct of the study.
* Bedridden patients.
* Presence of clinically unstable severe cardiovascular disease.
* Presence of clinically significant severe renal, hepatic or respiratory disease.
* Infection or dermatological condition at the proposed injection sites.
* Previous or planned participation in another clinical study (including the lower limb spasticity study of GSK1358820) within 6 months prior to the start of double-blind phase (Visit 2).
* Others whom the investigator or sub investigator considers not eligible for the study.
* Clinically significant severe reduction of muscle strength.
* Angle closure glaucoma or its preposition (narrow angle).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamaguchi

REFERENCES:
- [Derived] Kaji R, Osako Y, Suyama K, Maeda T, Uechi Y, Iwasaki M; GSK1358820 Spasticity Study Group. Botulinum toxin type A in post-stroke upper limb spasticity. Curr Med Res Opin. 2010 Aug;26(8):1983-92. doi: 10.1185/03007995.2010.497103. PMID 20569068

RESULTS

PARTICIPANT FLOW:
Groups:
- High-Dose BTX: BTX (GSK1358820) 200U (4 mL) was injected into the wrist and finger muscles, and 40U (0.8 mL) into the thumb muscles if thumb spasticity was present in the 12-week double-blind phase (DB) (once at Week 0)
- High-Dose Placebo: Placebo 4 mL was injected into the wrist and finger muscles, and 0.8 mL into the thumb muscles if thumb spasticity was present in the 12-week double-blind phase (DB) (once at Week 0)
- Low-Dose BTX: BTX (GSK1358820) 120U (2.4 mL) was injected into the wrist and finger muscles, and 30U (0.6 mL) into the thumb muscles if thumb spasticity was present in double-blind phase in the 12-week (DB) (once at Week 0)
- Low-Dose Placebo: Placebo 2.4 mL was injected into the wrist and finger muscles, and 0.6 mL into the thumb muscles if thumb spasticity was present in the 12-week double-blind phase (DB) (once at Week 0)
- DB High-Dose BTX + OL High-Dose BTX: BTX (GSK1358820) 200U (4 mL) was injected into the wrist and finger muscles, and 40U (0.8 mL) into the thumb muscles if thumb spasticity was present in the 12-week double-blind phase (DB) (once at Week 0) plus the 36-week open-label phase (OL) following the DB phase (up to 3 times, from Week 12 to Week 36 if participant met re-injection criteria [Modified Ashworth Scale (MAS) score of wrist >=2 and at least 12 weeks (84 days) since the last injection])
- DB High-Dose Placebo + OL High-Dose BTX: Placebo 4 mL was injected into the wrist and finger muscles, and 0.8 mL into the thumb muscles if thumb spasticity was present in the 12-week double-blind phase (DB) (once at Week 0) plus high-dose BTX in open-label phase (OL) following the DB phase (up to 3 times, from Week 12 to Week 36 if participant met re-injection criteria [Modified Ashworth Scale (MAS) score of wrist >=2 and at least 12 weeks (84 days) since the last injection])
- DB Low-Dose BTX + OL High-Dose BTX: BTX (GSK1358820) 120U (2.4 mL) was injected into the wrist and finger muscles, and 30U (0.6 mL) into the thumb muscles if thumb spasticity was present in double-blind phase in the 12-week (DB) (once at Week 0) plus high-dose BTX in open-label phase (OL) following the DB phase (up to 3 times, from Week 12 to Week 36 if participant met re-injection criteria [Modified Ashworth Scale (MAS) score of wrist >=2 and at least 12 weeks (84 days) since the last injection])
- DB Low-Dose Placebo + OL High-Dose BTX: Placebo 2.4 mL was injected into the wrist and finger muscles, and 0.6 mL into the thumb muscles if thumb spasticity was present in the 12-week double-blind phase (DB) (once at Week 0) plus high-dose BTX in open-label phase (OL) following the DB phase (up to 3 times, from Week 12 to Week 36 if participant met re-injection criteria [Modified Ashworth Scale (MAS) score of wrist >=2 and at least 12 weeks (84 days) since the last injection])
Period: Double-Blind Phase (12 Weeks)
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Started | 51 | 26 | 21 | 11 | 0 | 0 | 0 | 0
Completed | 47 | 25 | 21 | 11 | 0 | 0 | 0 | 0
Not Completed | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Phase (36 Weeks)
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Started | 0 | 0 | 0 | 0 | 47 | 25 | 21 | 11
Completed | 0 | 0 | 0 | 0 | 38 | 19 | 19 | 11
Not Completed | 0 | 0 | 0 | 0 | 9 | 6 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3 | 5 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0
Not completed — Concentrate on Treatment of Diabetes | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo | Total
Number analyzed (Participants) | 51 | 26 | 21 | 11 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.32) | 63.6 (11.03) | 62.7 (9.74) | 62.3 (9.61) | 63.2 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 2 | 6 | 35
  Male | 36 | 14 | 19 | 5 | 74
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese | 51 | 26 | 21 | 11 | 109

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for the Change From Baseline in Modified Ashworth Scale (MAS) Wrist Score to the End of the DB Phase (Week 12) in the High-dose Groups
Description: Change from baseline in MAS wrist score using a 6-point scale (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension) to each time point in the DB phase was calculated. In the graph plotting time points on the horizontal axis and changes from baseline on the vertical axis, the area surrounded by the MAS wrist score change curve and the horizontal axis was calculated and used as a summary index (AUC) for assessment of the MAS wrist score. Negative changes from baseline indicate improvement, and the AUC has a negative sign.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS): all participants randomized, with the exception of those who did not receive any investigational product and those with no assessment of post-treatment MAS wrist score
Measure: Mean (Standard Deviation); unit: Score*week
Arm/Group | High-Dose BTX | High-Dose Placebo
Number analyzed (Participants) | 51 | 26
Score*week | -10.397 (8.9313) | -3.567 (4.7189)
Statistical Analysis 1: Comparison: High-Dose BTX vs High-Dose Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -6.830, 95% CI [-10.567 to -3.093]

2. Secondary Outcome: Area Under the Curve (AUC) for the Change From Baseline in Modified Ashworth Scale (MAS) Wrist Score to the End of the DB Phase (Week 12) in the Low-dose Groups
Description: Change from baseline in MAS wrist score using a 6-point scale (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension) to each time point in the DB phase was calculated. In the graph plotting time points on the horizontal axis (HA) and changes from baseline on the vertical axis, the area surrounded by the MAS wrist score change curve and the HA was calculated and used as a summary index (AUC) for assessment of the MAS wrist score. Negative changes from baseline indicate improvement, and the area under the AUC has a negative sign.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score*week
Arm/Group | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 21 | 11
Score*week | -10.036 (7.7743) | -6.227 (8.6584)

3. Secondary Outcome: Mean Change From Baseline in MAS Wrist Score From Baseline to Week 12 of the Double-blind Phase
Description: The investigator assessed MAS wrist score using a 6-point scale (0, 1, 1+, 2, 3, and 4; 0=No increase in muscle tone to 4=Affected part[s] rigid in flexion or extension) at each time point in the double-blind phase. The "+1" (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder [less than half] of ROM [range of motion]) of MAS score is regarded as score 1.5.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | -0.66 (0.745) | -0.23 (0.430) | -0.86 (0.777) | -0.50 (0.742)
  Week 4 | -1.05 (0.912) | -0.48 (0.671) | -0.88 (0.740) | -0.73 (1.009)
  Week 6 | -1.15 (0.931) | -0.29 (0.569) | -0.95 (0.789) | -0.68 (0.956)
  Week 8 | -1.01 (0.970) | -0.35 (0.599) | -0.93 (0.884) | -0.50 (0.742)
  Week 12 | -0.83 (0.842) | -0.20 (0.408) | -0.71 (0.845) | -0.27 (0.647)

4. Secondary Outcome: Mean Change From Baseline in MAS Finger Score From Baseline to Week 12 of the Double-blind Phase
Description: The investigator assessed MAS finger score using a 6-point scale (0, 1, 1+, 2, 3, and 4; 0=No increase in muscle tone to 4=Affected part[s] rigid in flexion or extension) at each time point in the double-blind phase. The "+1" (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder [less than half] of ROM [range of motion]) of MAS score is regarded as score 1.5.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | -0.60 (0.671) | -0.19 (0.402) | -0.69 (0.733) | -0.23 (0.684)
  Week 4 | -0.92 (0.821) | -0.37 (0.657) | -0.95 (0.757) | -0.55 (0.688)
  Week 6 | -0.97 (0.800) | -0.33 (0.734) | -0.98 (0.782) | -0.23 (0.684)
  Week 8 | -0.86 (0.790) | -0.35 (0.759) | -0.69 (0.750) | -0.27 (0.518)
  Week 12 | -0.67 (0.709) | -0.26 (0.597) | -0.45 (0.947) | -0.14 (0.323)

5. Secondary Outcome: Mean Change From Baseline in Disability Assessment Scale (DAS) Score of Principal Measure From Baseline to Week 12 of the Double-blind Phase
Description: DAS scores of Hygiene, Pain, Dressing, and Limb posture were assessed using a 4-point scale (0=No functional disability to 3=Severe disability). Prior to the first injection, the investigator, in consultation with the participant, selected one functional disability item and assessed it as a principal measure at each time point in the double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | -0.49 (0.612) | -0.15 (0.368) | -0.67 (0.658) | 0.00 (0.000)
  Week 4 | -0.82 (0.748) | -0.31 (0.618) | -0.67 (0.577) | 0.00 (0.000)
  Week 6 | -0.86 (0.764) | -0.35 (0.629) | -0.67 (0.577) | -0.09 (0.302)
  Week 8 | -0.79 (0.771) | -0.38 (0.647) | -0.71 (0.561) | 0.00 (0.447)
  Week 12 | -0.70 (0.689) | -0.32 (0.557) | -0.57 (0.598) | 0.09 (0.302)

6. Secondary Outcome: Mean Change From Baseline in Disability Assessment Scale (DAS) Score of Hygiene From Baseline to week12 of the Double-blind Phase
Description: DAS score of Hygiene was assessed using a 4-point scale (0=No functional disability to 3=Severe disability) at each time point in double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | -0.27 (0.532) | -0.12 (0.431) | -0.43 (0.746) | -0.18 (0.405)
  Week 4 | -0.39 (0.603) | -0.23 (0.587) | -0.38 (0.669) | -0.36 (0.674)
  Week 6 | -0.43 (0.612) | -0.31 (0.618) | -0.43 (0.746) | -0.27 (0.467)
  Week 8 | -0.40 (0.676) | -0.29 (0.624) | -0.43 (0.746) | -0.18 (0.405)
  Week 12 | -0.34 (0.600) | -0.28 (0.678) | -0.33 (0.658) | -0.09 (0.539)

7. Secondary Outcome: Mean Change From Baseline in Disability Assessment Scale (DAS) Score of Pain From Baseline to Week 12 of the Double-blind Phase
Description: DAS score of pain was assessed using a 4-point scale (0=No functional disability to 3=Severe disability) at each time point in the double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | -0.10 (0.608) | 0.04 (0.344) | -0.14 (0.359) | 0.00 (0.000)
  Week 4 | -0.20 (0.749) | 0.04 (0.445) | -0.10 (0.436) | 0.00 (0.000)
  Week 6 | -0.20 (0.676) | -0.12 (0.588) | -0.10 (0.436) | -0.09 (0.302)
  Week 8 | -0.19 (0.673) | -0.04 (0.751) | -0.14 (0.478) | -0.09 (0.302)
  Week 12 | -0.09 (0.747) | 0.00 (0.645) | -0.14 (0.359) | -0.18 (0.405)

8. Secondary Outcome: Mean Change From Baseline in Disability Assessment Scale (DAS) Score of Dressing From Baseline to Week 12 of the Double-blind Phase
Description: DAS score of Dressing was assessed using a 4-point scale (0=No functional disability to 3=Severe disability) at each time point in the double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | -0.24 (0.586) | -0.04 (0.344) | -0.24 (0.436) | 0.00 (0.000)
  Week 4 | -0.24 (0.687) | 0.04 (0.662) | -0.33 (0.483) | 0.00 (0.000)
  Week 6 | -0.27 (0.785) | 0.04 (0.662) | -0.24 (0.436) | -0.09 (0.302)
  Week 8 | -0.21 (0.713) | 0.08 (0.717) | -0.38 (0.498) | -0.09 (0.302)
  Week 12 | -0.23 (0.633) | 0.12 (0.600) | -0.24 (0.436) | 0.00 (0.000)

9. Secondary Outcome: Mean Change From Baseline in Disability Assessment Scale (DAS) Score of Limb Posture From Baseline to Week 12 of the Double-blind Phase
Description: DAS score of Limb Posture was assessed using a 4-point scale (0=No functional disability to 3=Severe disability) at each time point in the double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | -0.43 (0.539) | -0.15 (0.368) | -0.33 (0.483) | -0.09 (0.302)
  Week 4 | -0.62 (0.602) | -0.12 (0.326) | -0.48 (0.602) | -0.09 (0.302)
  Week 6 | -0.69 (0.683) | -0.15 (0.464) | -0.67 (0.796) | -0.09 (0.302)
  Week 8 | -0.67 (0.694) | -0.21 (0.509) | -0.52 (0.680) | 0.00 (0.447)
  Week 12 | -0.57 (0.651) | -0.16 (0.473) | -0.43 (0.811) | -0.09 (0.539)

10. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Investigator From Baseline to Week 12 of the Double-blind Phase
Description: The CGI score of functional disability was assessed at each visit using the 11-point Numeric Rating Scale (NRS) (-5=Worst Possible to 5=Best Possible) at each time point in the double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | 1.14 (1.132) | 0.31 (0.838) | 0.86 (0.854) | 0.91 (1.044)
  Week 4 | 1.80 (1.456) | 0.50 (1.175) | 1.10 (1.044) | 0.45 (0.820)
  Week 6 | 1.61 (1.935) | 0.54 (1.208) | 1.00 (1.049) | 0.27 (0.905)
  Week 8 | 1.33 (1.950) | 0.42 (1.139) | 0.86 (1.108) | 0.27 (0.905)
  Week 12 | 0.94 (1.949) | 0.32 (1.108) | 0.10 (1.300) | 0.00 (0.894)

11. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Participant From Baseline to Week 12 of the Double-blind Phase
Description: as for outcome 10
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | 1.14 (1.296) | 0.73 (1.343) | 1.29 (1.231) | 0.36 (1.120)
  Week 4 | 1.53 (1.793) | 0.65 (1.938) | 1.48 (1.167) | 0.45 (2.252)
  Week 6 | 1.78 (1.918) | 0.73 (1.614) | 1.24 (1.411) | 0.55 (2.382)
  Week 8 | 1.52 (1.571) | 0.54 (1.318) | 1.19 (1.250) | 0.64 (2.461)
  Week 12 | 1.32 (1.733) | 0.92 (1.956) | 0.90 (1.136) | 0.18 (2.442)

12. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Physiotherapist/Occupational Therapist From Baseline to Week 12 of the Double-blind Phase
Description: as for outcome 10
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo
Number analyzed (Participants) | 51 | 26 | 21 | 11
Points on a scale
  Week 1 | 0.69 (0.860) | 0.46 (1.067) | 0.67 (0.730) | 0.36 (0.809)
  Week 4 | 1.08 (1.510) | 0.62 (1.203) | 0.86 (1.014) | 0.45 (0.934)
  Week 6 | 1.29 (1.683) | 0.62 (1.061) | 0.76 (1.300) | 0.27 (0.647)
  Week 8 | 0.98 (1.436) | 0.63 (0.970) | 0.71 (1.231) | 0.45 (1.036)
  Week 12 | 0.74 (1.421) | 0.64 (0.995) | 0.62 (1.359) | 0.36 (1.433)

13. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the MAS Wrist Score at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The investigator assessed the MAS wrist score using a 6-point scale (0, 1, 1+, 2, 3, and 4; 0=no increase in muscle tone to 4=affected part[s] rigid in flexion or extension) at each time point from baseline (at the start of the double-blind phase) to week 48. The "+1" (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder ([less than half] of ROM [range of motion]) of MAS score is regarded as score 1.5.
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | -1.53 (0.876) | -1.30 (0.849) | -1.53 (0.754) | -1.41 (0.437)
  Week 8 after first injection in OL | -1.30 (0.927) | -1.35 (0.922) | -1.53 (0.831) | -1.59 (0.801)
  Week 12 after first injection in OL | -1.07 (0.894) | -1.02 (0.858) | -1.11 (0.884) | -1.23 (0.984)
  Week 4 after second injection in OL | -1.61 (0.892) | -1.92 (0.943) | -1.34 (0.790) | -1.69 (0.530)
  Week 8 after second injection in OL | -1.41 (0.897) | -1.53 (0.882) | -1.34 (0.747) | -1.56 (0.563)
  Week 12 after second injection in OL | -1.03 (0.856) | -1.29 (0.751) | -1.09 (0.688) | -1.25 (0.707)
  Week 4 after third injection in OL | -1.36 (0.551) | -1.68 (0.405) | -1.17 (0.829) | -1.86 (0.690)
  Week 8 after third injection in OL | -1.28 (0.786) | -1.64 (0.505) | -1.28 (0.833) | -1.86 (0.627)
  Week 12 after third injection in OL | -1.18 (0.847) | -1.36 (0.636) | -1.06 (0.768) | -1.71 (0.488)

14. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the MAS Finger Score From at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The investigator assessed the MAS finger score using a 6-point scale (0, 1, 1+, 2, 3, and 4; 0=No increase in muscle tone to 4=Affected part[s] rigid in flexion or extension) at each time point from baseline (at the start of the double-blind phase) to week 48. The "+1" (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder [less than half] of ROM [range of motion]) of MAS score is regarded as score 1.5.
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | -1.21 (0.648) | -1.22 (0.850) | -1.26 (0.714) | -1.32 (0.603)
  Week 8 after first injection in OL | -1.14 (0.675) | -1.20 (0.938) | -1.08 (0.974) | -1.00 (0.742)
  Week 12 after first injection in OL | -0.89 (0.668) | -0.88 (0.757) | -0.92 (0.809) | -0.77 (0.720)
  Week 4 after second injection in OL | -1.40 (0.651) | -1.53 (0.675) | -1.19 (0.772) | -1.25 (0.463)
  Week 8 after second injection in OL | -1.06 (0.726) | -1.33 (0.748) | -1.16 (0.724) | -1.19 (0.704)
  Week 12 after second injection in OL | 0.89 (0.798) | -1.12 (1.024) | -1.00 (0.658) | -0.88 (0.641)
  Week 4 after third injection in OL | -1.36 (0.744) | -1.18 (0.751) | -1.44 (0.950) | -1.43 (0.673)
  Week 8 after third injection in OL | -1.20 (0.696) | -1.00 (1.072) | -1.28 (1.034) | -1.36 (0.476)
  Week 12 after third injection in OL | -1.03 (0.803) | -0.95 (0.961) | -1.28 (0.870) | -1.29 (0.699)

15. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Disability Assessment Scale (DAS) Score of Principal Measure at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: DAS scores of Hygiene, Pain, Dressing, and Limb posture were assessed using a 4-point scale (0=No functional disability to 3=Severe disability). Prior to the first injection, the investigator, in consultation with the participant, selected one functional disability item and assessed it as a principal measure at each time point from baseline (at the start of the double-blind phase) to Week 48.
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | -0.95 (0.785) | -0.96 (0.878) | -1.00 (0.882) | -0.64 (0.674)
  Week 8 after first injection in OL | -0.91 (0.718) | -0.96 (0.878) | -1.11 (0.832) | -0.73 (0.647)
  Week 12 after first injection in OL | -0.74 (0.734) | -0.86 (0.964) | -1.00 (0.767) | -0.64 (0.674)
  Week 4 after second injection in OL | -1.03 (0.707) | -1.39 (0.698) | -1.25 (0.931) | -0.88 (0.641)
  Week 8 after second injection in OL | -0.91 (0.712) | -1.33 (0.686) | -1.31 (0.946) | -0.88 (0.641)
  Week 12 after second injection in OL | -0.79 (0.740) | -1.41 (0.618) | -1.31 (0.873) | -0.88 (0.641)
  Week 4 after third injection in OL | -1.00 (0.548) | -1.18 (0.405) | -1.11 (0.782) | -0.71 (0.756)
  Week 8 after third injection in OL | -1.00 (0.562) | -1.18 (0.405) | -1.00 (0.866) | -0.71 (0.756)
  Week 12 after third injection in OL | -0.90 (0.553) | -1.09 (0.539) | -1.00 (0.707) | -0.86 (0.690)

16. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Disability Assessment Scale (DAS) Score of Hygiene at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The DAS score of Hygiene was assessed using a 4-point scale (0=No functional disability; 3=Severe disability) at each time point from baseline (at the start of the double-blind phase) to Week 48. BTX was injected in participants up to 3 times from Week 12 to Week 36 when participants met re-injection criteria. Measurements were taken at each point until Week 48 and summarized by the number of weeks after the re-injection in individuals (4, 8, and 12 weeks after each injection) in open-label phase; thus, measurements could have been taken up to Week 48 (12 weeks after the Week 36 injection).
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | -0.53 (0.767) | -0.83 (0.937) | -0.74 (0.806) | -0.45 (0.688)
  Week 8 after first injection in OL | -0.58 (0.731) | -0.70 (0.974) | -0.61 (0.850) | -0.55 (0.688)
  Week 12 after first injection in OL | -0.45 (0.705) | -0.62 (0.973) | -0.61 (0.850) | -0.55 (0.688)
  Week 4 after second injection in OL | -0.74 (0.780) | -0.83 (0.857) | -0.81 (0.981) | -0.38 (0.518)
  Week 8 after second injection in OL | -0.76 (0.781) | -0.83 (0.857) | -0.81 (0.981) | -0.38 (0.518)
  Week 12 after second injection in OL | -0.67 (0.816) | -0.82 (0.883) | -0.88 (0.957) | -0.25 (0.463)
  Week 4 after third injection in OL | -0.71 (0.644) | -0.55 (0.522) | -0.56 (0.726) | -0.14 (0.378)
  Week 8 after third injection in OL | -0.65 (0.587) | -0.55 (0.522) | -0.22 (0.972) | -0.29 (0.488)
  Week 12 after third injection in OL | -0.55 (0.510) | -0.45 (0.522) | -0.56 (0.726) | -0.29 (0.488)

17. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Disability Assessment Scale (DAS) Score of Pain at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The DAS score of Pain was assessed using a 4-point scale (0=No functional disability to 3=Severe disability) at each time point from baseline (at the start of the double-blind phase) to Week 48. BTX was injected in participants up to 3 times from Week 12 to Week 36 when participants met re-injection criteria. Measurements were taken at each point until Week 48 and summarized by the number of weeks after the re-injection in individuals (4, 8, and 12 weeks after each injection) in open-label phase; thus, measurements could have been taken up to Week 48 (12 weeks after the Week 36 injection).
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | -0.23 (0.527) | -0.22 (0.422) | -0.16 (0.501) | -0.27 (0.467)
  Week 8 after first injection in OL | -0.21 (0.559) | -0.22 (0.422) | -0.28 (0.669) | -0.18 (0.603)
  Week 12 after first injection in OL | -0.19 (0.594) | -0.24 (0.436) | -0.28 (0.575) | -0.27 (0.467)
  Week 4 after second injection in OL | -0.31 (0.718) | -0.22 (0.428) | -0.31 (0.704) | -0.13 (0.354)
  Week 8 after second injection in OL | -0.21 (0.592) | -0.28 (0.461) | -0.38 (0.719) | -0.25 (0.463)
  Week 12 after second injection in OL | -0.15 (0.508) | -0.29 (0.470) | -0.31 (0.704) | 0.00 (0.535)
  Week 4 after third injection in OL | -0.14 (0.478) | -0.18 (0.405) | -0.33 (0.707) | -0.14 (0.378)
  Week 8 after third injection in OL | -0.10 (0.447) | -0.18 (0.405) | -0.33 (0.707) | -0.29 (0.488)
  Week 12 after third injection in OL | -0.05 (0.510) | -0.09 (0.302) | -0.33 (0.707) | -0.29 (0.488)

18. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Disability Assessment Scale (DAS) Score of Dressing at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The DAS score of Dressing was assessed using a 4-point scale (0=No functional disability to 3=Severe disability) at each time point from baseline (at the start of the double-blind phase) to Week 48. BTX was injected in participants up to 3 times from Week 12 to Week 36 when participants met re-injection criteria. Measurements were taken at each point until Week 48 and summarized by the number of weeks after the re-injection in individuals (4, 8, and 12 weeks after each injection) in open-label phase; thus, measurements could have been taken up to Week 48 (12 weeks after the Week 36 injection).
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | -0.42 (0.763) | -0.13 (0.815) | -0.42 (0.507) | -0.27 (0.467)
  Week 8 after first injection in OL | -0.42 (0.731) | -0.30 (0.822) | -0.50 (0.514) | -0.36 (0.505)
  Week 12 after first injection in OL | -0.40 (0.767) | -0.19 (0.873) | -0.50 (0.514) | -0.36 (0.505)
  Week 4 after second injection in OL | -0.46 (0.701) | -0.39 (1.037) | -0.63 (0.500) | -0.50 (0.535)
  Week 8 after second injection in OL | -0.50 (0.749) | -0.28 (1.018) | -0.81 (0.655) | -0.50 (0.535)
  Week 12 after second injection in OL | -0.52 (0.755) | -0.35 (1.057) | -0.75 (0.447) | -0.50 (0.535)
  Week 4 after third injection in OL | -0.48 (0.680) | -0.55 (0.820) | -0.67 (0.500) | -0.43 (0.535)
  Week 8 after third injection in OL | -0.45 (0.686) | -0.64 (0.809) | -0.67 (0.500) | -0.43 (0.535)
  Week 12 after third injection in OL | -0.40 (0.681) | -0.45 (0.820) | -0.78 (0.441) | -0.57 (0.535)

19. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Disability Assessment Scale (DAS) Score of Limb Posture at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The DAS score of Limb Posture was assessed using a 4-point scale (0=No functional disability to 3=Severe disability) at each time point from baseline (at the start of the double-blind phase) to Week 48. BTX was injected in participants up to 3 times from Weeks 12 to 36 when participants met re-injection criteria. Measurements were taken at each point until Week 48 and summarized by the number of weeks after the re-injection in individuals (4, 8, and 12 weeks after each injection) in open-label phase; thus, measurements could have been taken up to Week 48 (12 weeks after the Week 36 injection).
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | -0.84 (0.843) | -0.74 (0.619) | -0.84 (0.834) | -0.73 (0.647)
  Week 8 after first injection in OL | -0.81 (0.764) | -0.74 (0.752) | -0.89 (0.758) | -0.73 (0.647)
  Week 12 after first injection in OL | -0.67 (0.786) | -0.67 (0.796) | -0.89 (0.832) | -0.64 (0.674)
  Week 4 after second injection in OL | -0.80 (0.677) | -1.00 (0.767) | -0.88 (0.806) | -0.75 (0.707)
  Week 8 after second injection in OL | -0.71 (0.719) | -1.06 (0.639) | -1.00 (0.816) | -0.75 (0.707)
  Week 12 after second injection in OL | -0.64 (0.742) | -1.12 (0.600) | -0.88 (0.806) | -0.75 (0.707)
  Week 4 after third injection in OL | -0.81 (0.602) | -1.00 (0.447) | -0.89 (0.782) | -0.57 (0.787)
  Week 8 after third injection in OL | -0.80 (0.616) | -1.00 (0.447) | -0.89 (0.782) | -0.71 (0.756)
  Week 12 after third injection in OL | -0.70 (0.733) | -0.91 (0.539) | -0.89 (0.601) | -0.71 (0.756)

20. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Investigator at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The CGI score of functional disability was assessed at each visit using the 11-point Numeric Rating Scale (NRS) (-5=Worst Possible to 5=Best Possible) at each time point from baseline (at the start of the double-blind phase) to Week 48.
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | 2.00 (2.000) | 1.83 (1.403) | 1.21 (1.548) | 1.36 (1.629)
  Week 8 after first injection in OL | 1.93 (2.005) | 1.83 (1.466) | 1.11 (1.641) | 1.73 (1.679)
  Week 12 after first injection in OL | 1.71 (1.979) | 1.71 (1.347) | 0.78 (1.957) | 1.09 (1.514)
  Week 4 after second injection in OL | 2.29 (2.163) | 2.78 (1.957) | 1.13 (1.708) | 2.38 (2.134)
  Week 8 after second injection in OL | 1.91 (2.094) | 2.67 (1.782) | 1.13 (1.586) | 2.25 (2.121)
  Week 12 after second injection in OL | 1.61 (2.030) | 2.29 (1.724) | 0.56 (1.825) | 1.88 (2.167)
  Week 4 after third injection in OL | 2.86 (1.682) | 2.55 (1.214) | 1.00 (1.000) | 2.86 (2.410)
  Week 8 after third injection in OL | 2.55 (1.791) | 2.82 (1.888) | 1.00 (1.000) | 3.14 (2.410)
  Week 12 after third injection in OL | 2.20 (1.735) | 2.00 (1.612) | 1.11 (1.054) | 2.71 (2.289)

21. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Participant at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: as for outcome 20
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | 1.60 (2.060) | 2.00 (2.045) | 1.79 (1.228) | 0.64 (2.580)
  Week 8 after first injection in OL | 1.79 (2.366) | 2.17 (2.188) | 1.83 (1.295) | 0.64 (2.656)
  Week 12 after first injection in OL | 1.79 (2.203) | 2.05 (1.962) | 1.67 (1.188) | 0.45 (2.583)
  Week 4 after second injection in OL | 2.00 (2.210) | 2.56 (2.770) | 2.06 (1.389) | 1.25 (3.536)
  Week 8 after second injection in OL | 1.91 (2.050) | 2.39 (2.831) | 1.88 (1.204) | 1.38 (3.583)
  Week 12 after second injection in OL | 1.88 (2.088) | 2.29 (2.616) | 1.88 (1.258) | 0.88 (3.399)
  Week 4 after third injection in OL | 2.76 (1.546) | 3.09 (1.700) | 2.22 (1.202) | 2.71 (2.812)
  Week 8 after third injection in OL | 2.90 (1.447) | 3.36 (1.912) | 2.44 (1.130) | 2.86 (2.410)
  Week 12 after third injection in OL | 2.70 (1.593) | 2.55 (2.162) | 2.11 (1.269) | 2.57 (2.573)

22. Secondary Outcome: Mean Change From Baseline (at the Start of the DB Phase) in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Physiotherapist/Occupational Therapist at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: as for outcome 20
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Number analyzed (Participants) | 43 | 23 | 20 | 11
Points on a scale
  Week 4 after first injection in OL | 1.37 (1.196) | 1.78 (1.204) | 0.95 (1.224) | 1.91 (2.343)
  Week 8 after first injection in OL | 1.47 (1.470) | 1.70 (1.222) | 0.94 (1.731) | 0.73 (0.786)
  Week 12 after first injection in OL | 1.29 (1.330) | 1.43 (1.207) | 1.33 (1.680) | 0.82 (1.662)
  Week 4 after second injection in OL | 1.74 (1.067) | 2.28 (1.965) | 1.69 (1.778) | 2.00 (1.512)
  Week 8 after second injection in OL | 1.56 (1.260) | 2.06 (1.924) | 1.25 (1.000) | 1.75 (1.282)
  Week 12 after second injection in OL | 1.36 (1.194) | 1.71 (1.490) | 1.00 (1.211) | 1.88 (2.167)
  Week 4 after third injection in OL | 1.90 (1.513) | 1.45 (1.036) | 1.00 (2.062) | 2.43 (1.134)
  Week 8 after third injection in OL | 1.30 (1.261) | 1.91 (1.973) | 1.89 (1.453) | 2.43 (1.512)
  Week 12 after third injection in OL | 1.20 (1.508) | 1.00 (1.414) | 1.78 (1.563) | 2.29 (1.704)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were classified by onset time because the study consists of the double-blind (DB) and open-label (OL) phases.
Description: AEs in the double-blind (DB) phase (Arms 1-4), AEs occurring after the start (injection) of the DB phase (Week 0), but before the first injection day in the open-label (OL) phase; AEs in the OL phase (Arms 5-8), AEs occurring after the first injection day in the OL phase. SAEs and AEs were analyzed in the Full Analysis Set.
Arm/Group | High-Dose BTX | High-Dose Placebo | Low-Dose BTX | Low-Dose Placebo | DB High-Dose BTX + OL High-Dose BTX | DB High-Dose Placebo + OL High-Dose BTX | DB Low-Dose BTX + OL High-Dose BTX | DB Low-Dose Placebo + OL High-Dose BTX
Serious Adverse Events (participants affected / at risk) | 6/51 | 3/26 | 1/21 | 0/11 | 4/43 | 3/23 | 4/20 | 0/11
Other Adverse Events (participants affected / at risk) | 17/51 | 12/26 | 8/21 | 6/11 | 21/43 | 12/23 | 14/20 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-Dose BTX (N=51) | High-Dose Placebo (N=26) | Low-Dose BTX (N=21) | Low-Dose Placebo (N=11) | DB High-Dose BTX + OL High-Dose BTX (N=43) | DB High-Dose Placebo + OL High-Dose BTX (N=23) | DB Low-Dose BTX + OL High-Dose BTX (N=20) | DB Low-Dose Placebo + OL High-Dose BTX (N=11)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic intracranial hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyothorax (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-Dose BTX (N=51) | High-Dose Placebo (N=26) | Low-Dose BTX (N=21) | Low-Dose Placebo (N=11) | DB High-Dose BTX + OL High-Dose BTX (N=43) | DB High-Dose Placebo + OL High-Dose BTX (N=23) | DB Low-Dose BTX + OL High-Dose BTX (N=20) | DB Low-Dose Placebo + OL High-Dose BTX (N=11)
Nasopharyngitis (Infections and infestations) | 7 | 4 | 3 | 1 | 8 | 3 | 5 | 5
Herpes zoster (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 1 | 4 | 2 | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Nail tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Frostbite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Edema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Grip strength decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exsanguination (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound hemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Posthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The frequency threshold (5%) for reporting other adverse events is based on the result of the double-blind phase for the first four arms listed in the table and on the open-label phase for the last four arms listed in the table.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.